CLINICAL TRIAL: NCT01473563
Title: Home Delivery of Pemetrexed as Maintenance Treatment in Patients Who Have Not Progressed After Induction Therapy for Advanced Nonsquamous Nonsmall Cell Lung Cancer: A Feasibility Study
Brief Title: A Study of Home Administration of Pemetrexed as Maintenance Treatment for Advanced Nonsquamous Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14079; H3E-EW-S133 (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Nonsquamous Non-Small Cell Neoplasm of Lung; Non-Small Cell Lung Cancer Metastatic; Non-Small Cell Lung Cancer Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): 500 milligrams per square meter (mg/m^2) pemetrexed administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Maintenance therapy administered until disease progression or the participant is discontinued for any other reason. The first dose of maintenance therapy will be administered at the hospital; thereafter, therapy will be administered in the home setting by qualified oncology homecare nurses.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Administered intravenously
  Other Names: LY231514; Alimta; Pemetrexed disodium; Pemetrexed sodium hydrate

SUMMARY:
The main purpose for this study is to answer the following research questions:

* Can pemetrexed be administered safely at the participant's home, using the same treatment procedure as in a hospital setting?
* Will the participant be satisfied with home care?
* How might this impact the participant's quality of life?
* What are the required medical resources needed to give pemetrexed in a home setting?

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of NSCLC defined as nonsquamous cell histology. Squamous cell and/or small cell histology is not permitted. Mixed NSCLC tumors will be categorized by the predominant cell type. NSCLC tumors that are not otherwise specified with regard to histology or cannot be subclassified as squamous, adenocarcinoma, or large cell histology will be categorized as nonsquamous
* Have Stage IIIB (not amenable to curative treatment) or Stage IV NSCLC prior to induction therapy as defined by the American Joint Committee on Cancer (AJCC) Staging Criteria for Lung Cancer
* Have completed 4 induction cycles of platinum-based doublet therapy (type at the discretion of the physician) for treatment of their advanced disease.
* Have not progressed after 4 cycles of induction therapy. Documented radiographic evidence of a tumor response must occur at the end of Cycle 4 of induction therapy within 3 weeks before receiving the first cycle of study drug [see Response Evaluation Criteria in Solid Tumors (RECIST), version (v) 1.1]
* Receive on-study treatment no earlier than 21 days and no later than 42 days from Cycle 4 Day 1 of induction therapy
* Have a Performance Status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Meet the following guidelines if the participant has received prior radiation therapy:

  * Previous radiation therapy is allowed to <25% of the bone marrow, but should have been limited and must not have included whole pelvis radiation
  * Participants must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia)
  * Participants who received palliative chest (in other words, thoracic skeleton including dorsal spine) or palliative extrathoracic radiotherapy to preexisting lesions are allowed to be enrolled in this trial
* Have adequate organ function, including:

  * Adequate bone marrow reserve: absolute neutrophil count (ANC) (segmented and bands) >=1.5x109/Liter (L), platelets >=100x109/L, and hemoglobin >=9 grams per deciliter (g/dL)
  * Hepatic: bilirubin <=1.5 x upper limit of normal (ULN) and alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) <=3.0 x ULN (ALP, AST, and ALT <=5.0 x ULN are acceptable if the liver has tumor involvement
  * Renal: calculated creatinine clearance (CrCl) >=45 milliliters per minute (mL/min) based on the original weight-based Cockcroft and Gault formula
* Are willing to comply with the following contraceptive criteria:

  * Females must be surgically sterile, postmenopausal or must have a negative serum or urine pregnancy test within 7 days prior to the first dose of study drug
  * Males and females with reproductive potential: Must agree to use a reliable method of birth control during the study and for 6 months following the last dose of study drug
* Have an estimated life expectancy of at least 12 weeks
* Have given written informed consent/assent prior to any study-specific procedures
* Are willing to comply with home delivery administration and have family or close environment support willing to comply with home delivery administration

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or no approved use of a drug or device (other than pemetrexed used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study
* Have a serious concomitant systemic disorder (for example, active infection including human immunodeficiency virus)
* Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants for at least 1 week before starting study treatment and their disease is asymptomatic and radiographically stable
* Are receiving concurrent administration of any other antitumor therapy
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results
* Are unable to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than aspirin dose ≤1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
* Are unable or unwilling to take folic acid or vitamin B12 supplementation
* Are unable or unwilling to take corticosteroids
* Are pregnant or lactating
* Have received a recent (within 30 days of enrollment) or are receiving concurrent yellow fever vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna
- United Kingdom (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maidstone, Kent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester, United Kingdom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huddersfield, West Yorkshire

REFERENCES:
- [Derived] Lal R, Bourayou N, Hillerdal G, Nicolson M, Vikstrom A, Lorenzo M, D'yachkova Y, Barriga S, Visseren-Grul C. Home administration of maintenance pemetrexed for patients with advanced non-squamous non-small cell lung cancer: rationale, practicalities and phase II feasibility study design. Health Qual Life Outcomes. 2013 Oct 3;11:163. doi: 10.1186/1477-7525-11-163. PMID 24090033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed study treatment and follow-up (FU) were considered to have completed the study. Participants received treatment until disease progression or discontinuation and were followed post treatment (post tx) discontinuation for up to 6 months.
Groups:
- Pemetrexed: Pemetrexed: 500 milligrams per meter squared (mg/m^2) administered as an intravenous (IV) infusion over approximately 10 minutes on Day 1 of each 21-day cycle until disease progression or the participant discontinued for any other reason. The first dose of maintenance therapy was administered at the hospital; thereafter, therapy was administered in the home setting by qualified oncology homecare nurses.
Period: Overall Study
Arm/Group | Pemetrexed
Started | 52
Received at Least 1 Dose of Study Drug | 52
Completed | 51
Not Completed | 1
Not completed — Lost to FU post tx discontinuation | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: Participants who received at least 1 dose of study drug.
Groups:
- Pemetrexed: Pemetrexed: 500 mg/m^2 IV infusion over approximately 10 minutes on Day 1 of each 21-day cycle until disease progression or the participant discontinued for any other reason. The first dose of maintenance therapy was administered at the hospital; thereafter, therapy was administered in the home setting by qualified oncology homecare nurses.
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 66.0 (12.05) [27.0 to 82.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 48
  Black or African American | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 43
  Sweden | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classified participants according to their functional impairment. Scores could have ranged from 0 (Fully Active) to 5 (Death).
  participants
    0: Fully Active | 14
    1: Restricted | 38
Most Recent Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma, Lung | 48
  Adenocarcinoma, Mucinous, No Other Symptoms (NOS) | 1
  Adenocarcinoma, Moderately Differentiated, Lung | 1
  Carcinoma, Non-Small Cell, Lung NOS | 2
Basis for Most Recent Pathological Diagnosis [Number; unit: participants]
  Cytological | 10
  Histopathological | 42
Stage of Disease [Number; unit: participants] — Disease stage described using American Joint Committee on Cancer (AJCC). Stages ranged from I (cancer was small and had not spread to the lymph nodes) to IV (cancer spread throughout the body). Stage III (cancer had spread to nearby tissue or lymph nodes) was further differentiated based on regional lymph nodes: Stage IIIA (spread to nearby lymph nodes) and Stage IIIB (spread to distance lymph nodes). The participant with Stage IIIA disease was enrolled in study because investigator considered participant not eligible for curative treatment.
  participants
    Stage IIIB | 3
    Stage IV | 48
    Stage IIIA | 1
Prior Systemic Therapy [Number; unit: participants] — Prior systemic therapies include carboplatin and gemcitabine; carboplatin and pemetrexed; cisplatin and pemetrexed; platinum-based therapy and pemetrexed. Participants pre-exposed to cisplatin and carboplatin were considered to have platinum-based therapy.
  participants
    Carboplatin + Gemcitabine | 9
    Carboplatin + Pemetrexed | 19
    Cisplatin + Pemetrexed | 20
    Platinum-Based Therapy + Pemetrexed | 4
Best Response to Prior Systemic Therapy [Number; unit: participants] — Best response to prior systemic therapy was defined using Response Evaluation Criteria In Solid Tumors [RECIST, version (v) 1.1] criteria. PR was having at least a 30% decrease in sum of longest diameter of target lesions; PD was having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir; SD was small changes that did not meet above criteria. Participant with PD (borderline tumor increase) was considered a protocol violation.
  participants
    Partial Response (PR) | 25
    Stable Disease (SD) | 26
    Progressive Disease (PD) | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Adhered to Treatment Administration at Home
Description: Participants were considered adherent from the time of the first dose in Cycle 1 (hospital administration) until either the last day of the cycle when the participant reverted to pemetrexed hospital administration or the last day of the cycle when the participant discontinued study treatment or the study for reasons related to the home setting. The percentage of participants who adhered to treatment administration at home was estimated by a Kaplan-Meier survival analyses approach. Participants who died or discontinued the study and treatment without reverting to hospital administration were censored at the time of discontinuation.
Time Frame: Cycle 1, Day 1 through Cycle 19, Day 1 and Cycle 19, Day 1 (21 days/cycle)
Population: Intention-to-Treat (ITT) population: Participants who received at least 1 dose of study drug. The number of participants censored was 6, 9, 7, 8, 7, 1, 0, 2, 2, 2, 2, 0, 3, 0, 0, 0, 0, 0, and 1 for Cycles 1 through 19, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
percentage of participants
  Cycle 1, Hospital Delivery | 100 [100 to 100]
  Cycle 2, Home Delivery | 98.0 [86.4 to 99.7]
  Cycle 3, Home Delivery | 98.0 [86.4 to 99.7]
  Cycle 4, Home Delivery | 98.0 [86.4 to 99.7]
  Cycle 5, Home Delivery | 98.0 [86.4 to 99.7]
  Cycle 6, Home Delivery | 98.0 [86.4 to 99.7]
  Cycle 7, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 8, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 9, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 10, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 11, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 12, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 13, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 14, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 15, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 16, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 17, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 18, Home Delivery | 90.7 [61.7 to 98.1]
  Cycle 19, Home Delivery | 90.7 [61.7 to 98.1]

2. Secondary Outcome: Change From Baseline in the European Quality of Life Instrument (EQ-5D) Visual Analogue Scale (VAS)
Description: The EQ-5D scale was used to provide an estimate of the health state utility in this population. The EQ-5D scale includes a 5-dimensional descriptive system that measures each of the health state attributes: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression according to a 3-point scale (no problem, some problems, and major problems) and a VAS that allows participants to rate their present health condition from 0 (worst imaginable health state) to 100 (best imaginable health state). The change from baseline in EQ-5D VAS is reported.
Time Frame: Baseline, Day 1 of Cycles 2 and 4 (21 days/cycle) and 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline EQ-5D VAS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed
Number analyzed (Participants) | 34
units on a scale
  Cycle 2 (n=34) | 3.0 (18.6)
  Cycle 4 (n=20) | 7.7 (21.7)
  30 days post treatment discontinuation (n=22) | -0.9 (18.9)

3. Secondary Outcome: Change From Baseline in the EQ-5D Index Score
Description: The EQ-5D scale was used to provide an estimate of the health state utility in this population. The EQ-5D scale includes a 5-dimensional descriptive system that measures each of the health state attributes: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression according to a 3-point scale (no problem, some problems, and major problems) and a VAS that allows participants to rate their present health condition from 0 (worst imaginable health state) to 100 (best imaginable health state). The change from baseline EQ-5D Index score is reported and the EQ-5D Index score was calculated by converting health state scores into a weighted health state index according to a United Kingdom population-based algorithm. The possible values for the EQ-5D Index score range from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension), on a scale where 1 represents the best possible health state.
Time Frame: Baseline, Day 1 of Cycles 2 and 4 (21 days/cycle) and 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline EQ-5D index assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed
Number analyzed (Participants) | 38
units on a scale
  Cycle 2 (n=38) | 0.03 (0.22)
  Cycle 4 (n=23) | 0.08 (0.22)
  30 days post treatment discontinuation (n=26) | -0.9 (0.28)

4. Secondary Outcome: Maximum Improvement Over Baseline in Individual Lung Cancer Symptoms Scale (LCSS) Item Scores
Description: LCSS is a 9-item questionnaire; 6 items are symptom-specific measures for lung cancer (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain), and 3 summation items describe overall symptomatic distress, interference with activity level, and overall quality of life during the past 24 hours. Participant responses were measured using a VAS with 100-millimeter (mm) lines. Scores ranged from 0 mm (no symptoms and no impact on activities, quality of life) to 100 mm (symptoms as bad as they could be, impacting activities and quality of life).
Time Frame: Baseline, Day 1 of each cycle (up to Cycle 19, 21 days/cycle), and 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline LCSS assessment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pemetrexed
Number analyzed (Participants) | 43
mm
  Loss of Appetite (n=43) | 16.3 (22.0)
  Fatigue (n=43) | 24.5 (27.2)
  Cough (n=41) | 9.2 (19.7)
  Dyspnea (n=41) | 17.2 (26.7)
  Hemoptysis (n=43) | 0.4 (4.3)
  Pain (n=40) | 11.8 (25.1)
  Overall Symptomatic Distress (n=43) | 8.3 (22.3)
  Interference With Activity Level (n=43) | 15.3 (25.1)
  Overall Quality of Life (n=41) | 12.2 (23.0)

5. Secondary Outcome: Participant Satisfaction: Chemotherapy at Hospital
Description: Participants were asked to evaluate their hospital experiences in this study by answering 4 questions (Q). Q1: "What do you consider advantages of having chemotherapy at the hospital? Choose all that apply." Choices included: "Support from other patients", "Access to other medical specialists", "Access to more technical services", "Safer in case something goes wrong", and "Other". Q2: "What do you consider disadvantages of having chemotherapy at the hospital? Choose all that apply." Choices included: "Need to travel", "Having to wait for treatment", "Not having a personalized treatment", "Lack of privacy on the ward", and "Other". Q3: "How would you rate your overall satisfaction with chemotherapy at the hospital?" and Q4: "How would you rate your overall satisfaction with the nursing staff during chemotherapy at the hospital?" Choices for Q3 and Q4 included: "Very dissatisfied", "Somewhat dissatisfied", "Neither satisfied nor dissatisfied", "Somewhat satisfied", or "Very satisfied".
Time Frame: The first evaluation completed at either Cycle 4, Day 1 (21 days/cycle) or 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and answered at least 1 of the specified questions.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 39
participants
  Q1, Support from other patients | 8
  Q1, Access to other medical specialists | 19
  Q1, Access to more technical services | 12
  Q1, Safer in case something goes wrong | 19
  Q1, Other | 3
  Q2, Need to travel | 36
  Q2, Having to wait for treatment | 27
  Q2, Not having a personalized treatment | 5
  Q2, Lack of privacy on the ward | 7
  Q2, Other | 1
  Q3, Very dissatisfied | 0
  Q3, Somewhat dissatisfied | 3
  Q3, Neither satisfied nor dissatisfied | 3
  Q3, Somewhat satisfied | 11
  Q3, Very satisfied | 21
  Q4, Very dissatisfied | 3
  Q4, Somewhat dissatisfied | 0
  Q4, Neither satisfied nor dissatisfied | 0
  Q4, Somewhat satisfied | 3
  Q4, Very satisfied | 32

6. Secondary Outcome: Participant Satisfaction: Chemotherapy at Home
Description: Participants were asked to evaluate their home treatment experiences in this study by answering 4 questions (Q). Q5: "What do you do consider advantages of having chemotherapy at home? Choose all that apply." Choices included: "No need to travel", "Not having to wait for treatment", "Personalized service", "More privacy", and "Other". Q6:"What do you consider disadvantages of having chemotherapy at home? Choose all that apply." Choices included: "Lack of other patients' support", "Extra burden for family/friends", "Safety concerns", "Need to rely on 1 medical specialist", and "Other". Q7: "How would you rate your overall satisfaction with chemotherapy at home?" Choices included: "Very dissatisfied", "Somewhat dissatisfied", "Neither satisfied nor dissatisfied", "Somewhat satisfied", or "Very satisfied".
Time Frame: The first evaluation completed at either Cycle 4, Day 1 (21 days/cycle) or 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and answered at least 1 of the specified questions.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 39
participants
  Q5, No need to travel | 37
  Q5, Not having to wait for treatment | 27
  Q5, Personalized service | 28
  Q5, More privacy | 20
  Q5, Other | 2
  Q6, Lack of other patients' support | 5
  Q6, Extra burden for family/friends | 1
  Q6, Safety concerns | 4
  Q6, Need to rely on 1 medical specialist | 7
  Q6, Other | 19
  Q7, Very dissatisfied | 1
  Q7, Somewhat dissatisfied | 0
  Q7, Neither satisfied nor dissatisfied | 2
  Q7, Somewhat satisfied | 1
  Q7, Very Satisfied | 30

7. Secondary Outcome: Participant Satisfaction: Regarding the Study Nurse
Description: Participants were asked 7 questions (Q) about their study nurse for home treatment. Q8: "Was the nurse an easy person to talk to?", Q9: "When the nurse came, did you feel he/she had enough time to do the required things?", Q10: "Do you think the nurse had time to discuss things with you?", Q11: "Did you feel that the nurse knew enough about you and your illness?" Choices for Q8 through Q11 included: "Yes" or "No". Q12: "Were you able to get all the information you wanted about your illness or treatment?" Choices included: "Yes", "No", or "Uncertain". Q13: "Would you say that the nurse gave…" Choices included: "a lot of reassurance and support", "some reassurance and support", or "hardly any reassurance and support". Q14: "How would you rate your overall satisfaction with the nursing staff during chemotherapy at home?" Choices included: "Very dissatisfied", "Somewhat dissatisfied", "Neither satisfied nor dissatisfied", "Somewhat satisfied", or "Very satisfied".
Time Frame: The first evaluation completed at either Cycle 4, Day 1 (21 days/cycle) or 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and answered at least 1 of the specified questions.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 38
participants
  Q8, Yes | 37
  Q8, No | 0
  Q9, Yes | 36
  Q9, No | 1
  Q10, Yes | 37
  Q10, No | 1
  Q11, Yes | 36
  Q11, No | 0
  Q12, Yes | 34
  Q12, No | 0
  Q12, Uncertain | 3
  Q13, Hardly any reassurance and support | 0
  Q13, Some reassurance and support | 2
  Q13, A lot of reassurance and support | 35
  Q14, Very dissatisfied | 3
  Q14, Somewhat dissatisfied | 0
  Q14, Neither satisfied nor dissatisfied | 1
  Q14, Somewhat satisfied | 1
  Q14, Very satisfied | 33

8. Secondary Outcome: Participant Satisfaction: Preferences Regarding Home and/or Hospital Treatment
Description: Participants were asked to evaluate their preferences regarding home and/or hospital treatment delivery in this study by answering 2 questions (Q). Q15: "Do you prefer having your chemotherapy at home or at the hospital, or are you indifferent?" Choices included: "Home", "Hospital", or "Indifferent". Q16: "Would you recommend having chemotherapy at home to someone else in your same situation?" Choices included: "Yes", "No", or "Not sure".
Time Frame: The first evaluation completed at either Cycle 4, Day 1 (21 days/cycle) or 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and answered at least 1 of the specified questions.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 38
participants
  Q15, Home | 33
  Q15, Hospital | 0
  Q15, Indifferent | 5
  Q16, Yes | 37
  Q16, No | 0
  Q16, Not sure | 0

9. Secondary Outcome: Physician Satisfaction: Distant Management of Participant
Description: The physician was asked, "How would you rate your overall satisfaction with the distant management of the participant during chemotherapy at home?" Choices included: "Very dissatisfied", "Somewhat dissatisfied", "Neither satisfied nor dissatisfied", "Somewhat satisfied", or "Very satisfied".
Time Frame: 30 days post treatment discontinuation
Population: Participants who received at least 1 dose of study drug and for whom the investigator answered the specified question at 30 days post treatment discontinuation.
Measure: Number; unit: investigators
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
investigators
  Very Dissatisfied | 2
  Somewhat Dissatisfied | 1
  Neither Satisfied Nor Dissatisfied | 0
  Somewhat Satisfied | 8
  Very Satisfied | 20

10. Secondary Outcome: Resource Utilization: Number of Participants With an Unplanned Use of Healthcare Resources
Description: The number of participants who had at least 1 unplanned use of health care resources [accident and emergency department (dept.), specialists [oncologist, pulmonologist, etcetera (etc.)], general practitioner (GP) or family doctor, or diagnostic procedures] during the study is reported.
Time Frame: Cycle 1, Day 1 through last day of cycle when participant reverted to hospital administration or discontinued (up to Cycle 19, 21 days/cycle)
Population: ITT population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
participants | 29

11. Secondary Outcome: Resource Utilization: Unplanned Health Care Visits, Consultations, and Diagnostic Services
Description: The unplanned use of any 1 of the following 4 resources is reported, as well as the unplanned use of each resource: accident and emergency dept., specialists (oncologist, pulmonologist etc.), GP or family doctor, and diagnostic procedures. Results are reported as the number of participants with an unplanned resource use (visit) for a specified number of times.
Time Frame: as for outcome 10
Population: Participants who received at least 1 dose of study drug and had at least 1 unplanned use of health care resources.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 29
participants
  1 Unplanned Visit, Any Resource | 8
  2 Unplanned Visits, Any Resource | 6
  3 Unplanned Visits, Any Resource | 5
  4 Unplanned Visits, Any Resource | 2
  5 Unplanned Visits, Any Resource | 3
  9 Unplanned Visits, Any Resource | 1
  10 Unplanned Visits, Any Resource | 1
  13 Unplanned Visits, Any Resource | 1
  1 Unplanned Visit, Accident and Emergency Dept. | 7
  2 Unplanned Visits, Accident and Emergency Dept. | 2
  3 Unplanned Visits, Accident and Emergency Dept. | 2
  1 Unplanned Visit, Specialist | 9
  2 Unplanned Visits, Specialist | 3
  5 Unplanned Visits, Specialist | 1
  1 Unplanned Visit, GP or Family Doctor | 6
  2 Unplanned Visits, GP or Family Doctor | 3
  3 Unplanned Visits, GP or Family Doctor | 2
  4 Unplanned Visits, GP or Family Doctor | 3
  1 Unplanned Visit, Diagnostic procedures | 6
  2 Unplanned Visits, Diagnostic procedures | 2
  3 Unplanned Visits, Diagnostic procedures | 3
  4 Unplanned Visits, Diagnostic procedures | 1

12. Other Pre Specified Outcome: Number of Participants Who Had Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), or Died
Description: The number of participants who had at least 1 TEAE or serious TEAE (regardless of causality) is reported along with the number of participants who died (due to any cause) while on therapy or during treatment discontinuation follow-up (up to 6 months). TEAEs started on or after the date and time of first dose of study drug, or started prior to study drug but worsened after study drug started. Clinically significant events were defined as SAEs and other non-serious adverse events (AEs). A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: First dose of study drug (Cycle 1, Day 1) through study completion [up to Cycle 19 (21 days/cycle) or treatment discontinuation, plus up to 6 months post treatment discontinuation]
Population: Safety Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
participants
  At least 1 TEAE | 51
  At least 1 Serious TEAE | 21
  Death, AE (fell, multiple injuries) | 1
  Death, Study Drug Toxicity (atypical pneumonia) | 1
  Death, Study Disease | 26

13. Secondary Outcome: Resource Utilization: Duration of Health Care Visits
Description: The duration of the health care visit in the home setting is reported. The visit started when the nurse arrived and included the entire treatment process. The visit ended when the nurse left the home setting. Due to the limited number of participants with evaluable data, results are reported for Cycles 2 through 4.
Time Frame: Cycle 2, Day 1 through last day of cycle when participant reverted to hospital administration or discontinued (up to Cycle 4, 21 days/cycle)
Population: Participants who received at least 1 dose of study drug and had at least 1 health care visit in the home setting from Cycle 2 through Cycle 4.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pemetrexed
Number analyzed (Participants) | 42
hours
  Cycle 2 (n=42) | 1.67 (0.493)
  Cycle 3 (n=35) | 1.66 (0.683)
  Cycle 4 (n=28) | 1.57 (0.311)

14. Secondary Outcome: Resource Utilization: Distances Traveled
Description: The distance traveled is reported by region (Great Britain and Sweden) and includes the distance traveled by the participant from his/her home to the hospital (Cycle 1) and other cycles where the homecare nurse traveled from the hospital to the participant's home. Due to the limited number of participants with evaluable data, results are reported for Cycles 1 through 4.
Time Frame: Cycle 1, Day 1 through last day of cycle when participant reverted to hospital administration or discontinued (up to Cycle 4, 21 days/cycle)
Population: Participants who received at least 1 dose of study drug and had data for distance traveled for at least 1 cycle from Cycle 1 through Cycle 4.
Measure: Mean (Standard Deviation); unit: kilometers (km)
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
kilometers (km)
  Cycle 1, Home to Hospital, Great Britain (n=25) | 19.7 (23.39)
  Cycle 1, Home to Hospital, Sweden (n=7) | 30.7 (23.08)
  Cycle 2, Hospital to Home, Great Britain (n=24) | 15.5 (13.12)
  Cycle 2, Hospital to Home, Sweden (n=7) | 23.9 (23.93)
  Cycle 3, Hospital to Home, Great Britain (n=11) | 23.8 (16.72)
  Cycle 3, Hospital to Home, Sweden (n=4) | 17.5 (17.97)
  Cycle 4, Hospital to Home, Great Britain (n=7) | 11.7 (8.75)
  Cycle 4, Hospital to Home, Sweden (n=2) | 24.5 (27.58)

15. Secondary Outcome: Overall Survival (OS) at 6 Months
Description: The percentage of participants who were alive at Month 6 was calculated as a cumulative percentage by Kaplan-Meier survival analyses approach. For participants not known to have died as of the cut-off date, OS was censored as the last contact date (known alive).
Time Frame: Cycle 1, Day 1 to the date of death from any cause (up to Month 6)
Population: ITT population: Participants who received at least 1 dose of study drug. Twenty-four (24) participants were censored (alive) at the end of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
percentage of participants | 73 [58.1 to 82.8]

16. Secondary Outcome: Time to Treatment Failure (TTF)
Description: The time from the date of the first dose of study treatment (Cycle 1, Day 1) to the date of death from any cause, PD (clinical and objective), or discontinuation of pemetrexed due to toxicity. Response was defined using RECIST, v1.1 criteria. PD was defined as having at least a 20% increase in the sum of the longest diameter of target lesions and at a minimum 5 mm increase above nadir. TTF was censored at the date of the last visit for participants who did not discontinue pemetrexed, who were still alive, and who had not progressed.
Time Frame: Cycle 1, Day 1 to first event (up to Cycle 19, 21 days/cycle)
Population: ITT population: Participants who received at least 1 dose of study drug. Two (2) participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 52
months | 3.0 [2.3 to 4.2]

ADVERSE EVENTS:
Time Frame: Baseline through study completion [up to Cycle 19 (21 days/cycle) or treatment discontinuation, plus up to 6 months post treatment discontinuation]
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 23/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=52)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Device occlusion (General disorders) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=52)
Anaemia (Blood and lymphatic system disorders) | 12 (14)
Lacrimation increased (Eye disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 17 (24)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (8)
Chest pain (General disorders) | 4 (4)
Fatigue (General disorders) | 20 (31)
Influenza like illness (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 3 (4)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (7)
Bronchitis (Infections and infestations) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Blood creatinine increased (Investigations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (11)
Lethargy (Nervous system disorders) | 9 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
A thorough literature search revealed that no specific validated questionnaire was available to assess participant and physician satisfaction with home care or resource utilization, therefore specific questions were created by the sponsor for use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days